CLINICAL TRIAL: NCT04086628
Title: Evaluation of the Immunization Coverage Against Influenza in Children With Asthma Followed at the Hospital of Nancy
Brief Title: Influenza Vaccine in Children With Asthma
Acronym: VAGA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A01944-53
Record Dates: First submitted 2019-08-22; First posted 2019-09-11 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Asthma in Children; Influenza Vaccine; Immunization Coverage
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthmatic children vaccinated
- Asthmatic children unvaccinated

SUMMARY:
The occurence of influenza can be a factor of imbalance of asthma. Asthma patients are recommended for annual influenza vaccination . However there is insufficient vaccination coverage of asthmatic patients despite this recommendation. The aim of this study is to evaluate the rate of influenza vaccination coverage of children with asthma aged from 6 month to 17 years of age followed in pediatric pneumology consultation at the university hospital of Nancy.

DETAILED DESCRIPTION:
Using a questionnaire, the investigator will estimate the percentage of the asthmatic patients vaccinated against influenza. He will then compare the 2 groups of vaccinated and unvaccinated patients : comparison of patients characteristics, comparison of asthma characteristics (severity, asthma control...). He will also analyze the causes of vaccination or non-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* asthmatic patients followed in pediatric pneumology consultation at university hospital of Nancy aged from 6 months to 17 years

Exclusion Criteria:

* asthmatic children who have been followed for less than 1 year

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with asthma
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of asthmatic patients vaccinated against influenza | through study completion, an average of 6 months
  Percentage of patients vaccinated against influenza will be evaluate among children with asthma followed in pediatric pneumology consultation.

SECONDARY OUTCOMES:
Socio-demographic characteristics of patients | through study completion, an average of 6 months
  Socio-demographic characteristics will be recorded from the questionnaire and compare between the 2 groups : vaccinated and unvaccinated patients.
Age of patients (years) | through study completion, an average of 6 months
  Age of patients will be recorded from the questionnaire and compared between the 2 groups : vaccinated and unvaccinated patients.
Asthma severity (mild, moderate, severe asthma) | through study completion, an average of 6 months
  Asthma severity (mild, moderate, severe asthma) is assessed from the level of treatment required to control symptoms according to Global Initiative for Asthma (GINA) 2018 recommendations. The investigator will compare asthma severity between the 2 groups : vaccinated and unvaccinated patients.
Asthma symptom control (well controled, partly controlled, uncontrolled) | through study completion, an average of 6 months
  Level of asthma symptoms control (well controled, partly controlled, uncontrolled) is assessed from symptoms control tool, according to GINA 2018 recommendations. The investigator will compare asthma symptom control between the 2 groups : vaccinated and unvaccinated patients.

CONTACTS AND LOCATIONS:
Overall Officials: Aurore Blondé, Dr, Principal Investigator — CHRU nancy
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No